CLINICAL TRIAL: NCT06694623
Title: Keratinized Tissue Regeneration Following Apically Positioned Flap with and Without Free Gingival Graft Strip: a Split Mouth Randomized Clinical Trial
Brief Title: Keratinized Tissue Gain Following Apically Positioned Flap with and Without Free Gingival Graft Strip
Acronym: FGGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adam Malesevic (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Sponsor-Investigator, Adam Malesevic, Associate professor, University of Novi Sad
Organization: University of Novi Sad (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 106/2-2023; Faculty of Dentistry Pancevo (Other: Faculty of Dentistry, Clinic for Oral surgery)
Record Dates: First submitted 2024-11-06; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Keratinized Mucosa
Keywords: keratinized mucosa; free gingival graft strip; apically positioned flap; wound contraction

STUDY DESIGN:
Intervention Model Description: Split mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- apically positioned flap alone (Active Comparator): apically positioned flap alone
  Interventions: Procedure: Apically positioned flap
- apically positioned flap with FGG strip (Active Comparator): apically positioned flap with FGG strip
  Interventions: Procedure: Apically positioned flap with FGG strip

INTERVENTIONS:
Procedure: Apically positioned flap — The split thickness flap was apically positioned as much as possible and sutured to the periosteum utilizing T-mattress sutures.
  Arms: apically positioned flap alone
Procedure: Apically positioned flap with FGG strip — The split thickness flap was apically positioned as much as possible and sutured to the periosteum utilizing T-mattress sutures. FGG strip was sutured to the apical end of recipient bed.
  Arms: apically positioned flap with FGG strip

SUMMARY:
In non-implant edentulous patients reduction of height and width of residual alveolar ridge and reduced attached KT compromise the denture-bearing area unambiguously leading to decrease in full denture stability and retention. Furthermore, in implant edentulous patients insufficient KT is associated with increased plaque accumulation, tissue inflammation, soft tissue recession, marginal bone loss and increased prevalence of peri-implantitis. The present study aimed to evaluate keratinized tissue gain and the wound contraction rate between apically positioned flap without and with free gingival graft strip over a 6-month follow up period.

This research was designed as split mouth controlled clinical study included 17 patients having edentulous upper jaw with reduced width of keratinized tissue ( ≤ 4mm measured from middle of the crest to the buccal mucogingival junction or ≤ 2mm from occluso-buccal edge of the alveolar ridge to the mucogingival junction). In each patient, both surgical techniques, apically positioned flap without and with free gingival graft strip, were applied simultaneously. The change of keratinized tissue width and wound contraction rate were measured 30, 60 , 90 and 180 days after surgery

DETAILED DESCRIPTION:
The surgical procedure was done by one experienced surgeon. Before surgery, patients were given to rinse the mouth with 0,12% clorhexidine gluconate for 1 minute. Following the local anesthesia utilizing Artikaine 4% with 1:100000 epinephrine the elevation of split-thickness flap was started. Incision was done at the level of MGJ from maxillary tuberosity on one side to tuberosity of the opposite side. Initially, sharp dissection was carefully done in an apical direction to leave exposed periosteum without tearing. Further, blunt dissection was used to advance periosteum exposure and muscle fibres detachment. For apically positioned flap group the split thickness flap was apically positioned as much as possible and sutured to the periosteum utilizing T-mattress sutures. Regarding free gingival graft strip group, after the split thickness flap was sutured apically, free gingival graft in the form of strip, harvested from the palate, was sutured to the apical end of the recipient bed leaving the rest of periosteum to heal by secondary epitelization. Free gingival graft strip stabilized with 6-0 resorbable sutures by means of two single interrupted and cross-mattress sutures. The dimensions of free gingival graft strip was 30-35mm in length (depending on the length of the apical part of recipient bed), 2-3mm in width and 1-1.5mm in thick. The palatal donor site was sutured using cross-mattress sutures. Patients were given postoperative instructions which included antibiotics regime (amoxicillin 500mg, 3x1 for 5 days or in case of penicillin allergy- clindamycin 600mg, 2x1 5 days) and rinsing with chlorehexidine solution 0.12% two times a day for 14 days.

To control for bias, measurements were carried out by one examiner not involved in the surgical procedure. Measurements were taken from regions representing tooth #16 to tooth #26. The colour-coded periodontal probe (University of North Caroline Probe CP15 PCPUNC156, Hy Friedy) utilized to measure the distance from depth of newly formed vestibule to the edge of vertical cut made on the GM representing position of certain tooth. Measurement for each tooth were summarized in three regions: anterior group (central and lateral incisor region)- AG, middle group (canine, first and second premolar region)- MG and posterior group (first molar region)- PG.

First measurement was done immediately after surgery (T0) and represented the distance from depth of newly formed vestibule to the edge of vertical cut made on the GM (for apically positioned flap group) and from apical margin of free gingival graft strip to the edge of vertical cut made on the GM (for free gingival graft strip group). Follow up measurements were taken at 30 (T1), 60 (T2) , 90 (T3) and 180 (T4) days after surgery.

Primary outcome was wound contraction rate representing the percentage of keratinized tissue reduction between time point immediately after surgery (T0, 100%) and follow-up time points (T1,T2,T3 and T4). Secondary outcomes were 1) patient-reported outcomes such as patient discomfort and pain which was evaluated utilizing visual analogue scale (VAS) at 1, 2, 7 and 10 days after surgery and the amount of ibuprofen taking within 10 days after surgery, 2) the surgery time which represented the time from first incision to the last suture with a digital timer rounded to the whole minutes, 3) wound infection (yes/no), and wound bleeding (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* patients with edentulous upper jaws which are not able to wear full upper denture owing to compromise retention and stability being 18 years old or older,
* patients with reduced width of keratinized tissue (≤ 4mm) measured from middle of the crest to the buccal mucogingival junction ( the distance from occluso-buccal edge of the alveolar ridge to the mucogingival junction ≤ 2mm), - patients who belong to ASA1 or ASA2, according to the American Academy to Anesthesiology
* patients who do not suffer from any systemic disease affecting wound healing,
* patients which are able to provide a signed informed consent and are able to comply with determined follow-up time points.

Exclusion Criteria:

* patient is a heavy smoker (more than 10 cigarettes per day),
* patients with history of malignancy, radiotherapy or chemotherapy within the 5 years,
* pregnant or nursing patients,
* patients who are taking medications which have an effect on mucosal healing in general (steroids, non-steroidal anti-inflammatory drugs taken in high doses and in long term, bisphosphonates).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Wound contraction rate | From enrollment to the 180 day
  Percentage of tissue tissue contraction during healing period

SECONDARY OUTCOMES:
Pain | 1, 2, 7 and 10 day postoperatively
  Visual Analogue Scale (VAS) 100mm long will be used. The greater the value the greater the pain. The left end of scale is 0mm (no pain), and the right end of scale iz 100mm (the greatest pain that patient can imagine).
number of ibuprofen tablets | 1, 2, 7, 10 days postoperatively
Surgery duration | From start to the end of surgery
  Duration of surgery will be recorded in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Pancevo, Pančevo, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urban IA, Lozada JL, Nagy K, Sanz M. Treatment of severe mucogingival defects with a combination of strip gingival grafts and a xenogeneic collagen matrix: a prospective case series study. Int J Periodontics Restorative Dent. 2015 May-Jun;35(3):345-53. doi: 10.11607/prd.2287. PMID 25909521
- [Background] Arnoux JP, Papasotiriou A, Weisgold AS. A revised technique for stage-two surgery in the severely resorbed mandible: a technical note. Int J Oral Maxillofac Implants. 1998 Jul-Aug;13(4):565-8. PMID 9714965
- [Background] Gamal N, Shemais N, Al-Nawawy M, Ghallab NA. Post-extraction volumetric analysis of alveolar ridge contour using subepithelial connective tissue graft in esthetic zone: a randomized controlled clinical trial. Clin Oral Investig. 2023 Nov;27(11):6503-6512. doi: 10.1007/s00784-023-05255-0. Epub 2023 Sep 19. PMID 37726486
- [Background] Song YW, Yoon SW, Cha JK, Jung UW, Jung RE, Thoma DS. Soft Tissue Dimensions Following Tooth Extraction in the Posterior Maxilla: A Randomized Clinical Trial Comparing Alveolar Ridge Preservation to Spontaneous Healing. J Clin Med. 2020 Aug 10;9(8):2583. doi: 10.3390/jcm9082583. PMID 32784997
- [Background] De Angelis P, De Rosa G, Manicone PF, De Giorgi A, Cavalcanti C, Speranza A, Grassi R, D'Addona A. Hard and soft tissue evaluation of alveolar ridge preservation compared to spontaneous healing: a retrospective clinical and volumetric analysis. Int J Implant Dent. 2022 Dec 8;8(1):62. doi: 10.1186/s40729-022-00456-w. PMID 36480055
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475